CLINICAL TRIAL: NCT07047079
Title: The Effectiveness of a Patient-navigation-based Preoperative Rehabilitation Exercise Program in Patients Undergoing Total Knee Arthroplasty: A Randomised Controlled Trial
Brief Title: Patient-navigation-based Preoperative Rehabilitation Exercise Program in Patients Undergoing TKA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Sun (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other)
Responsible Party: Sponsor-Investigator, Anna Sun, Nurse Practitioner, First Affiliated Hospital of Jinan University
Organization: First Affiliated Hospital of Jinan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KY-2025-105
Record Dates: First submitted 2025-06-13; First posted 2025-07-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Total Knee Arthroplasty; Knee Osteoarthritis
Keywords: Patient navigation; Preoperative exercise; Total Knee Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autonomous preoperative rehabilitation exercise program (Other): Participants will receive an autonomous preoperative rehabilitation program from admission day to surgery day (preoperative).
  Interventions: Other: Autonomous preoperative rehabilitation exercises
- Patient-navigation-based preoperative rehabilitation exercise program (Other): Participants will receive a patient-navigation-based preoperative rehabilitation exercise programme from admission day to surgery day (preoperative).
  Interventions: Other: The navigator provided full-period preoperative rehabilitation exercise guidance+navigation services

INTERVENTIONS:
Other: Autonomous preoperative rehabilitation exercises — 1. Method: On the day of admission, a research assistant provided a verbal explanation of the preoperative rehabilitation exercise regimen and distributed a guidance manual. Participants are advised to perform self-directed exercises 2-3 times daily according to the manual from admission day to surgery day (preoperative). They were also advised to promptly inform ward medical staff of any unusual conditions or concerns.
  2. Preoperative rehabilitation exercise regimen:
     * Pulmonary function exercises: including abdominal breathing exercises and effective cough learning.
     * Quadriceps strength exercises: including straight leg raises and lateral leg raises.
     * Knee range of motion exercises: including knee flexion exercises and knee extension exercises.
     * Lower limb thrombosis prevention exercises: ankle pump exercise
  Arms: Autonomous preoperative rehabilitation exercise program
Other: The navigator provided full-period preoperative rehabilitation exercise guidance+navigation services — 1. The navigator's guidance preoperative rehabilitation exercise regimen was identical to that of the control group, but offered full-period guidance, including the following:
     1. On the day of admission, in addition to the same measures as the control group, the navigators demonstrated the exercise movements and required participants to perform return demonstrations to ensure mastery of the exercises.
     2. During the preoperative period, navigators conducted daily ward visits, offering two 20-minute supervised sessions and sending nightly exercise reminders between 7:00-8:00 PM.
  2. Navigation services covered seven areas:
  establishing contact with participants or carers, providing disease-related education, assessing needs and facilitating resources, offering social and emotional support, providing interpretation services upon request, identifying and resolving exercise barriers, and promoting self-management.
  Arms: Patient-navigation-based preoperative rehabilitation exercise program

SUMMARY:
This study aimed to assess the effectiveness of a patient navigation-based preoperative rehabilitation exercise program for patients undergoing total knee arthroplasty.

DETAILED DESCRIPTION:
Participants were recruited from among patients newly admitted to the orthopaedic ward who met the selection criteria. Participants who provided written informed consent completed a survey collecting demographic and clinical information, followed by a baseline assessment (T0). Subsequently, they were randomly assigned to either the control group or the experimental group. Participants in both groups received standardised, identical inpatient rehabilitation and nursing services throughout their hospitalisation. From admission day to surgery day (preoperative), control group participants will receive an autonomous preoperative rehabilitation exercise programme, while experimental group participants will receive a patient-navigation-based preoperative rehabilitation exercise programme

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with knee osteoarthritis (KOA) scheduled to undergo primary unilateral total knee arthroplasty (TKA)
* Assessed by the attending physician as medically fit to tolerate preoperative rehabilitation exercise, possessing effective communication skills, and capable of cooperating with all required examinations and assessments
* Assessed as capable (either the patient or their caregiver) of using a smartphone to receive information

Exclusion Criteria:

* Individuals unable to cooperate due to impaired consciousness, cognitive impairment, or similar conditions
* Concurrent severe comorbidities such as liver cirrhosis, respiratory failure, renal failure, malignant tumors, trauma, etc.
* History of significant neuromuscular disorders or other joint diseases deemed by the attending physician to affect joint function
* a time interval of greater than 7 days or less than 3 days between the admission day date and the scheduled surgery date;
* Currently undergoing systematic lower limb functional exercise training within the past four weeks

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
knee osteoarthritis severity | Outcome will be measured five times: hospital admission (baseline, T0), surgery day (preoperative) (T1),1 weeks after the operation (T2),2 weeks after the operation (T3),and 4 weeks after the operation (T4)
  Knee osteoarthritis severity will be measured using the Chinese version of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Scale. The scale consists of 24 items divided into three subscales: pain (5 items), stiffness (2 items), and physical function (17 items). Each item is scored on a scale of 0 to 4. The scores are recoded into a 96-point total scale, where higher scores indicate greater severity of knee osteoarthritis.

SECONDARY OUTCOMES:
Exercise adherence | Outcome will be measured five times: hospital admission (baseline, T0), surgery day (preoperative) (T1),1 weeks after the operation (T2),2 weeks after the operation (T3),and 4 weeks after the operation (T4)
  The exercise adherence was measured using the Orthopaedic Patient Functional Exercise Compliance Scale, developed by Chinese scholars. This scale comprises three components: adherence to physical exercises (8 items), adherence to psychological exercises (4 items), and adherence to active learning exercises (3 items). Each item is scored using a 5-point Likert scale, where 1 point indicates "not at all able to do it" and 5 points indicate "completely able to do it". Higher scores represent better adherence.
Self-efficacy | Outcome will be measured five times: hospital admission (baseline, T0), surgery day (preoperative) (T1),1 weeks after the operation (T2),2 weeks after the operation (T3),and 4 weeks after the operation (T4)
  Self-efficacy was measured using the Chinese version of the Self-Efficacy for Rehabilitation Outcome Scale.This scale is designed to measure patients' belief in their ability to perform behaviours typical of physical rehabilitation for knee surgery. It comprises two sections, totaling 12 items: Rehabilitation Exercise Self-Efficacy (5 items) and Coping Self-Efficacy (7 items). Each item is rated using an 11-point Likert scale, where 0 indicates "Cannot do at all" and 10 indicates "Can do without any difficulty". The total score is 120. Higher scores indicate stronger rehabilitation self-efficacy beliefs in the patient.
Knee joint function | Outcome will be measured five times: hospital admission (baseline, T0), surgery day (preoperative) (T1),1 weeks after the operation (T2),2 weeks after the operation (T3),and 4 weeks after the operation (T4)
  Knee joint function will be measured using the Hospital for Special Surgery (HSS) Knee Scoring System. This scale comprises seven sections. This 100-point scoring system includes pain (30 points), function (22 points), range of motion (18 points, one point per eight degrees), muscle strength (10 points), flexion deformity (10 points), and stability (10 points). Points are deducted if patients use walking aids or present with flexion contracture or varus/valgus deformities. Total scores range from 0 to 100, with higher values reflecting superior knee joint function.
Knee range of motion (ROM) | Outcome will be measured five times: hospital admission (baseline, T0), surgery day (preoperative) (T1),1 weeks after the operation (T2),2 weeks after the operation (T3),and 4 weeks after the operation (T4)
  Knee range of motion (ROM) will be measured with a goniometer. The normal ROM values for the knee joint are as follows: flexion from 0° to 135°, extension to 0° (with some individuals exhibiting hyperextension ranging from 0° to 10°). The active range of motion (AROM) spans from 0° to 135°, while the passive range of motion (PROM) can reach up to 150°.
Pain intensity | Outcome will be measured five times: hospital admission (baseline, T0), surgery day (preoperative) (T1),1 weeks after the operation (T2),2 weeks after the operation (T3),and 4 weeks after the operation (T4)
  Pain intensity will be measured using the Visual Analogue Scale (VAS). The VAS consists of a 10-centimetre horizontal line divided into 10 equal intervals, where higher scores represent greater pain intensity. A score of 0 denotes no pain, whereas a score of 10 denotes the most severe pain imaginable. Patients are instructed to mark the point on the line corresponding to their perceived pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sun, Principal Investigator — research team
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT07047079/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/79/NCT07047079/ICF_001.pdf